CLINICAL TRIAL: NCT01728337
Title: Phase IV, Randomized, Double-blind Study on Muscle Activity of Two Commercial Preparations of Botulinum Toxin Type A (Dysport and Xeomin) Administered to the Upper Third of the Face (Forehead Lines).
Brief Title: Phase IV Study On Muscle Activity Of Two Commercial Preparations Of Botulinum
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hexsel Dermatology Clinic (Other)
Responsible Party: Principal Investigator, Doris Hexsel, MD, Hexsel Dermatology Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12-2012
Record Dates: First submitted 2012-11-07; First posted 2012-11-19 (Estimated); Results first posted 2014-08-11 (Estimated); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Sun-induced Wrinkles
Keywords: botulinum toxin,; wrinkles
MeSH Terms: interventions — abobotulinumtoxinA; Botulinum Toxins, Type A; incobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dysport and Xeomin (Active Comparator): 30 U of Dysport® was injected on the right side of the forehead and 12 U Xeomin® was injected on the left side of the forehead (dose-equivalence 2.5:1).
  Interventions: Drug: Dysport; Drug: Xeomin
- Xeomin and Dysport (Active Comparator): 30 U Dysport® was injected on the left side of the forehead and 12 U Xeomin® was injected on the right side of the forehead (dose-equivalence 2.5:1).
  Interventions: Drug: Dysport; Drug: Xeomin

INTERVENTIONS:
Drug: Dysport — Dysport® was injected on the right side of the forehead and Xeomin® was injected on the left side of the forehead.
  Other Names: botulinum toxin type A
Drug: Xeomin — Xeomin® was injected on the right side of the forehead and Dysport® was injected on the left side of the forehead
  Other Names: botulinum toxin type A

SUMMARY:
this study was proposed to provide more scientific and objective data on the clinical and aesthetic effects of these two toxins (Dysport and Xeomin).

DETAILED DESCRIPTION:
Subjects will perform 6 (six) visits during the study:

Screening visit, performed 30 to 1 day before the visit 1, when eligible subjects will be recruited and first evaluations will be performed; visit 1, which is the baseline and when the injections will be performed; visit 2, 30 +/- 3 days after the injections, when evaluations will be performed; visit 3, 90 +/- 3 days after the injections, when evaluations will be performed; 4, 120 +/- 3 days after the injections, when evaluations will be performed; visit 5, 150 +/- 3 days after the injections, when evaluations will be performed.

Assessment of percentage (%) of responders, after 5 months of injection, to the effects of two BT-A preparations, Dysport® and Xeomin®, by measuring frontalis m. wrinkle intensity at maximum contraction, as measured by visual Wrinkles Severity Scale (WSS).

ELIGIBILITY:
Inclusion Criteria:

* Subject agreement to provide written informed consent and the willingness and ability to comply with all aspects of the protocol;
* Female subjects;
* Phototype I to IV;
* Subjects aged between 18 and 60 years;
* Subjects naive for BT-A treatment;
* Subjects presenting the same degree of moderate (2) to severe (3) wrinkles on the left and right side of forehead under maximum voluntary contraction of the frontalis m. according WSS;
* Subjects with Minor's test showing at least grade III in the Sweating Intensity Visual Scale;
* Medical history and physical examination which, based on the investigator's opinion, do not prevent the subject from taking part in the study or from making use of the products under investigation;
* Subjects of childbearing age should present a negative urine pregnancy test at baseline and should be using a highly effective contraceptive method during all study;
* Availability of the subject throughout the study (5 months);
* Subject agreeing not to undergo other cosmetic or dermatological procedures during the participation in the study;
* Subjects with sufficient schooling and knowledge to enable them to cooperate to the degree required by the protocol.

Exclusion Criteria:

* Pregnant women or women intending to become pregnant in the following 5 months after screening;
* Lactation period;
* Subjects participating in other clinical trials;
* Any prior surgery affecting the frontalis and/or orbicularis muscles, prior blepharoplasty or brow lift;
* Any prior cosmetic procedures, including fillers, or scars that may interfere with the study results;
* Subjects with neoplastic, muscular or neurological diseases;
* Subjects taking aminoglycoside and penicillamine antibiotics, quinine or Ca2+ channel blockers;
* Subjects with inflammation or active infection in the area to be injected;
* Subjects presenting evident facial asymmetry;
* Subjects with a history of adverse effects, such as sensitivity to the components of any of the study drug formula, ptosis or any other adverse effect which, in the investigator's opinion, should prevent the subject from participating in the study;
* Subjects presenting Myasthenia Gravis, Eaton-Lambert Syndrome and motor neuron disease;
* Subjects with coagulation disorders or taking anticoagulants;
* Subjects with known systemic autoimmune diseases;
* Subjects with a history of non-adherence to medical treatment or showing unwillingness to adhere to the study protocol;
* Any condition that, in the opinion of the investigator, can compromise the evaluation of the study.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2011-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Doris Hexsel, MD, Principal Investigator — Brazilian Center for Dermatologic Studies
Locations (1):
- Brazilian Center For Studies in Dermatology, Porto Alegre, Rio Grande do Sul, Brazil

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients included in this study were recruted from two research centers.
Pre-assignment Details: We did not have any drop-out in this study.
Groups:
- Dysport and Xeomin: Dysport® was injected on the one side of the forehead and Xeomin® was injected on the other side of the forehead.
Period: Overall Study
Arm/Group | Dysport and Xeomin
Started | 80
Completed | 80
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Xeomin and Dysport: Xeomin® was injected on the one side of the forehead and Dysport® was injected on the other side of the forehead.
Arm/Group | Xeomin and Dysport
Number analyzed (Participants) | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 80
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80
  Male | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 80
Evoked Compound Muscle Action Potentials [Mean (Standard Deviation); unit: mV] — The Evoked Compound Muscle Action Potentials (CMAP) is the sum of the action potentials of individual muscle fibers obtained by stimulating a motor nerve. It is obtained through a set surface electrode on the point of the motor muscle and a reference electrode placed on an electrically neutral area (usually on a tendon). The amplitude of the CMAP reflects the number of muscle fibers depolarized in response to a stimulus and is measured in millivolts (mV).
  mV | 1053 (282)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Responders After 5 Months After the Procedure
Description: Percentage (%) of responders, after 5 months of injection, to the effects of two botulinum toxin type A (BT-A), Dysport® and Xeomin®. Responders were defined as individuals who presented at least 1 score less in the Wrinkles Scale Score (WSS) at maximum contraction compared to the WSS score at baseline.
  WSS is a validated 4-point scale, at rest and at maximum voluntary contraction of the frontalis muscle, in which 0 means no wrinkles up to 3 which means sever wrinkles.
Time Frame: 5 months after intervention
Population: 80 sujbects were included in this study, each patient have received both products in their faces. The randomization was performed to define the side for each product.
Measure: Number; unit: percentage of participants
Arm/Group | Dysport | Xeomin
Number analyzed (Participants) | 80 | 80
percentage of participants | 37 | 34

2. Secondary Outcome: Maximum Evoked Compound Muscle Action Potential
Description: To evaluate the duration, magnitude and peak of effects of two BT-A preparations, by measuring of the maximum Evoked Compound Muscle Action Potentials after contraction.
Time Frame: 5 months after the procedure.
Population: All subjects have received both treatments.
Measure: Mean (Standard Deviation); unit: mV
Arm/Group | Dysport | Xeomin
Number analyzed (Participants) | 80 | 80
mV | 694 (391) | 677 (387)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Dysport | Xeomin
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/80
Other Adverse Events (participants affected / at risk) | 2/80 | 2/80
OTHER ADVERSE EVENTS (reported when occurring in more than 1.25% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dysport (N=80) | Xeomin (N=80)
Worsening of Glabellar frown lines (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — Worsening of Glabellar frown lines, transitory and related to the study medication.
Injection site bleeding (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — Injection site bleeding, not related to the study medication. It was associated to the injection.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No